CLINICAL TRIAL: NCT06935669
Title: Randomised Controlled Clinical Trial Analgesic Effect of Bupivacaine Plus Ketamine Versus Bupivacaine Alone in Transversalis Fascia Plane Block After Cesarean Section Under Spinal Anaesthesia
Brief Title: Analgesic Effect of Bupivacaine Plus Ketamine Versus Bupivacaine Alone in Transversalis Fascia Plane Block
Acronym: TFBP
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FMASU MD36/2025
Record Dates: First submitted 2025-04-04; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-03

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia | interventions — Ketamine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketamine and bupivacaine (Experimental): Transversalis fascia plane block
  Interventions: Drug: Ketamine; Drug: Bupivacain
- Bupivacaine alone (Active Comparator): Transversalis fascia plane block
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Ketamine — Patients in this group will receive a transversalis fascia plane block using a combination of bupivacaine and ketamine.
  Other Names: Ketalar
  Arms: Ketamine and bupivacaine
Drug: Bupivacaine — Control group to evaluate the additional effect of ketamine in the experimental arm.
  Other Names: Marcaine
  Arms: Bupivacaine alone
Drug: Bupivacain — Patients in this group will receive a transversalis fascia plane block using a combination of bupivacaine and ketamine.
  Other Names: Marcaine
  Arms: Ketamine and bupivacaine

SUMMARY:
The objective of this study is to compare the efficacy of transversalis fascia plane block using bupivacaine and ketamine versus bupivacaine alone for pain management after cesarean section under spinal anaesthesia.

DETAILED DESCRIPTION:
Cesarean section (CS) is one of the most common surgeries and usually causes moderate to severe pain for up to 48 h. The rate of CS, which is a life-saving surgical procedure in cases of certain complications that occur during pregnancy and birth, has exceeded 20% worldwide Pain control after CS has crucial importance, especially in the first 24 h, to facilitate early ambulation and the establishment of breastfeeding. Insufficient analgesia in the postoperative period may cause a number of undesirable effects, such as patient discomfort, thromboembolism due to extended immobilization, and increased pulmonary secretions resulting in complications The well-known side effects of analgesic morphine as nausea, vomiting, itching and sedation, may interfere with the interaction between mother and child, breastfeeding and post-partum experience in a dose-dependent manner. However, a number of alternative strategies have been described in order to reduce morphine consumption post-operatively .

The mode and type of analgesia should be safe and effective. A stimulus caused by a lesion in tissue or organs during surgery is the cause of postoperative pain .

The primary source of pain after abdominal surgeries, including CS, are the anterior abdominal wall and abdominal viscera, and blocking these areas could provide proper postoperative analgesia .

Recently, the application of fascial plane blocks has increased due to the widespread use of ultrasound among anesthesiologists and the avoidance of opioids in a multimodal analgesic strategy. Different regional anesthetic techniques have been introduced, including ilioinguinal nerve blocks, abdominal field blocks, Transversalis Fascia Plane (TFP) blocks, and Transversus Abdominis Plane (TAP) blocks to alleviate pain from the abdominal wall incision .

Transversalis Fascia Plane, performed in the posterior axillary line, blocks branches of L1 nerve roots, including ilioinguinal and iliohypogastric nerves. This method has been used to control postoperative pain in patients undergoing different lower abdominal surgeries A variety of anesthetic agents such as bupivacaine, levobupivacaine, and ropivacaine are commonly used in TAP blocks. These drugs provide short-term analgesia and primarily alleviate somatic pain. To extend the duration of analgesic efficacy, various adjuvants such as opioids, ketamine, clonidine, and alpha-2 agonists like dexmedetomidine have been added .

Bupivacaine is one of the widely used local analgesics. ketamine affects pain modulation through multiple mechanisms of action. It is a non-competitive N-methyl-d-aspartate (NMDA) receptor antagonist, which exerts an anti-hyperalgesic effect by decreasing central sensitization and reducing the wind-up phenomenon in the postoperative period .

The aim of this study is to investigate the effect of transversalis fascia plane block using bupivacaine plus ketamine on postoperative pain compared to bupivacaine alone in patients undergoing cesarean section under spinal anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients aging ≥ 21 years to ≤ 45.
* Patients undergoing cesarean section under spinal anesthesia.
* American Society of Anesthesiologists (ASA) physical statusphysical status classes II.

Exclusion Criteria:

* Patient's refusal of procedure or participation in the study.
* Coagulopathy and bleeding disorders.
* Use of chronic pain medications.
* Pregnancy-induced hypertension or diabetes.
* Evidence of Local skin infections at site of injection.
* Body mass index >40kg/m2
* A history of relevant local anesthetic allergy.

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-04-25 (Estimated); Primary Completion 2026-04-25 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
The mean VAS pain on movement will be recorded as the primary outcome of the study | day 1
  Pain intensity will be assessed using the Visual Analog Scale (VAS), where 0 = no pain and 10 = worst pain.
  Patients will report their pain levels at rest and during movement at 24 hours after the transversalis fascia plane block.
  The mean VAS score will be compared between the ketamine + bupivacaine group and the bupivacaine-only group.

SECONDARY OUTCOMES:
Time to first rescue analgesia will be recorded | Day 1
  Time (in minutes/hours) from the completion of the transversalis fascia plane block to the administration of the first dose of rescue analgesia will be recorded.
  Rescue analgesia will be given when the patient reports a VAS score ≥ 4 or requests additional pain relief.
  A longer time to first rescue analgesia in the ketamine + bupivacaine group would indicate prolonged analgesic duration compared to the bupivacaine-only group.
total requirements of rescue analgesia Nalbuphine over the first 24 hours postoperative will be recorded | Day 1
  Rescue analgesia will be given when the patient reports a VAS score ≥ 4 or requests additional pain relief.

CONTACTS AND LOCATIONS:
Overall Officials: AHMED Ad Elgamal, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University faculty of medicine, Cairo, Egypt, Egypt

REFERENCES:
- [Background] Hassan, Shamsul Kamaruljan, et al. "Comparison of analgesic efficacy and safety of bupivacaine plus ketamine versus bupivacaine alone in rectus sheath block for midline laparotomy." Anaesthesia, Pain & Intensive Care 27.2 (2023): 154-160.